CLINICAL TRIAL: NCT04501198
Title: Moxibustion Combined With Characteristic Lifestyle Intervention of Traditional Chinese Medicine in the Treatment of Abdominal Obesity: A Study Protocol for a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hubei Hospital of Traditional Chinese Medicine (Other)
Collaborators: Shanxi Provincial Hospital of Traditional Chinese Medicine (Unknown); Shenzhen Bao'an Traditional Chinese Medicine Hospital Group (Unknown); Wuhan Hospital of Traditional Chinese Medicine (Other); Xiangyang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Wang Jian, professor, Hubei Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202006009
Record Dates: First submitted 2020-07-23; First posted 2020-08-06 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Obesity
Keywords: abdominal obesity; moxibustion; characteristic lifestyle intervention
MeSH Terms: conditions — Obesity; Obesity, Abdominal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moxibustion with characteristic lifestyle intervention of TCM (Experimental): Participants will receive moxibustion combined with characteristic lifestyle intervention of traditional chinese medicine.In this study, xiusheng decoction, traditional exercises, and modern lifestyle intervention will be combined as the characteristic lifestyle intervention method of TCM to help participants establish healthy living habits. Participants will receive the treatment of moxibustion 6 times a week to fulfill a 8-session treatment course, and the intervention of Xiusheng Decoction and Traditional exercises will last for 8 weeks.While the intervention of modern lifestyle intervention will be conducted for 12 weeks including the treatment period of 8 weeks and the follow-up period of 4 weeks.
  Interventions: Device: moxibustion combined with characteristic lifestyle intervention of traditional chinese medicine
- moxibustion with lifestyle intervention (Experimental): Participants will receive moxibustion combined with lifestyle intervention. Participants will receive the treatment of moxibustion 6 times a week to fulfill a 8-session treatment course,while the intervention of modern lifestyle intervention will be conducted for 12 weeks including the treatment period of 8 weeks and the follow-up period of 4 weeks.
  Interventions: Device: Moxibustion combined with lifestyle intervention.
- lifestyle intervention (Other): Participants will receive lifestyle intervention which includes modern dietary exercise modifications. Participants will receive this treatment for a 8-session treatment course and 4-session follow-up course.
  Interventions: Device: lifestyle intervention

INTERVENTIONS:
Device: moxibustion combined with characteristic lifestyle intervention of traditional chinese medicine — 1. The moxibustion acupoints will be selected as①zhongwan, guanyuan, shenque, and zusanli;②pishu,shenshu. Acupoints group①will be selected on Monday, Wednesday, and Friday, Acupoints group②will be selected on Tuesday, Thursday, Saturday.Moxibustion treatment will be applied once every day, 6 times per week, for 8 consecutive weeks.
  2. Xiusheng decoction, traditional exercises, and modern lifestyle intervention will be combined as the characteristic lifestyle intervention method of TCM to help participants establish healthy living habits. The Xiusheng Decoction should be taken twice a day. Traditional exercises will be taken for 35~40 minutes everyday, 7 times a week. The intervention of Xiusheng Decoction and traditional exercises will be conducted for 8 weeks. All patients will be instructed to follow a good living habits which will last 12 weeks including the treatment period of 8 weeks and the follow-up period of 4 weeks.
  Arms: Moxibustion with characteristic lifestyle intervention of TCM
Device: Moxibustion combined with lifestyle intervention. — 1. The moxibustion acupoints will be selected as①zhongwan, guanyuan, shenque, and zusanli;②pishu,shenshu. Acupoints group①will be selected on Monday, Wednesday, and Friday, Acupoints group②will be selected on Tuesday, Thursday, Saturday.Moxibustion treatment will be applied once every day, 6 times per week, for 8 consecutive weeks.
  2. All patients will be instructed to follow a good living habits including diet and exercise intervention which will last 12 weeks including the treatment period of 8 weeks and the follow-up period of 4 weeks.
  Arms: moxibustion with lifestyle intervention
Device: lifestyle intervention — All patients will be instructed to follow a good living habits including diet and exercise intervention which will last 12 weeks including the treatment period of 8 weeks and the follow-up period of 4 weeks.
  Arms: lifestyle intervention

SUMMARY:
This study will investigate whether the combination of moxibustion and characteristic lifestyle intervention of TCM can alleviate the clinical symptoms and improve quality of life and mental health in patients with abdominal obesity. The results are expected to provide clinical evidence for the application of the combination of moxibustion and characteristic lifestyle intervention of TCM in patients with abdominal obesity.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial conducted from January, 2020 to January, 2022 that includes 150 participants who have abdominal obesity and meet the eligibility criteria. The participants will be randomly divided into 3 groups in a 2:2:1 allocation ratio.The intervention group will receive moxibustion combined with characteristic lifestyle intervention of TCM;the other group will receive moxibustion combined with lifestyle intervention;the control group will receive lifestyle intervention only.Each treatment will last 12 weeks including 8 weeks of intervention period and 4 weeks of follow-up period. The primary outcome is the waist circumference(WC),the secondary outcomes include obesity-related indicators,serum biochemical indexs,blood pressure, conversion score of constitution characteristics, and measurement of the scale.Adverse events will be recorded during the intervention and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Patients recruited for this study should meet the following inclusion criteria:

1.Satisfying the criteria for the diagnosis of abdominal obesity; 2.18 years old≤age≤55 years old; 3.Being able to fully understand and voluntarily sign informed consent.

Exclusion Criteria:

Patients with any of the following criteria will be excluded from the study:

1. Presence of endocrine disorders such as: polycystic ovary syndrome; Cushing's syndrome; uncorrected thyroid disease.
2. Presence of diabetes mellitus, or hypertension, or abnormal liver and kidney functions, or mental diseases.
3. Pregnant or lactating state, women who plan to become pregnant within 12 weeks.
4. History of bulimia, anorexia, or any other eating disorders.
5. Use of medications in the past 3 months, such as diet drugs, corticosteroids, antidepressants, which may affect weight or appetite.
6. History of surgical weight loss, postoperative adhesions.
7. History of participating in a clinical study of weight loss or any other therapies to lose weight in the past 3 months.
8. Presence of local skin rupture, allergy and scar constitution.
9. Unable to cooperate with the research caused by other diseases or reasons.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Changes in waistline | week 0,week 2,week 4,week 6,week 8,week 12
  Waist circumference will be measured around the abdomen at the level of the umbilicus (belly button).

SECONDARY OUTCOMES:
Changes in weight | week 0,week 2,week 4,week 6,week 8,week 12
  Body weight will be measured by a body composition analyzer (OMRON V.BODY).
Changes in body mass index | week 0,week 2,week 4,week 6,week 8,week 12
  Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Changes in body fat percentage | week 0,week 2,week 4,week 6,week 8,week 12
  The body fat percentage (BFP) of a human or other living being is the total mass of fat divided by total body mass, multiplied by 100. Body fat percentage will be measured by a body composition analyzer (OMRON V.BODY).
Changes in basal metabolic value | week 0,week 2,week 4,week 6,week 8,week 12
  Basal metabolic value will be measured by a body composition analyzer (OMRON V.BODY).
Changes in hip circumference | week 0,week 2,week 4,week 6,week 8,week 12
  hip circumference will be measured at the level of maximum posterior extension of the buttocks.
Changes in waist-to-hip circumference ratio | week 0,week 2,week 4,week 6,week 8,week 12
  waist-to-hip ratio is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement ( W ÷ H ).
Changes in fasting blood-glucose | week 0, week 8
  examined with the blood sample
Changes in fasting insulin | week 0, week 8
  examined with the blood sample
Changes in insulin resistance index insulin resistance index insulin resistance index | week 0, week 8
  examined with the blood sample
Changes in total cholesterol | week 0, week 8
  examined with the blood sample
Changes in triglyceride | week 0, week 8
  examined with the blood sample
Changes in low density lipoprotein | week 0, week 8
  examined with the blood sample
Changes in high-density lipoprotein | week 0, week 8
  examined with the blood sample
Changes in uric acid | week 0, week 8
  examined with the blood sample
Changes in blood pressure | week 0, week 8
  Both Systolic and diastolic blood pressure assessed by office and ambulatory blood pressure monitoring(mmHg).
Changes in Conversion score of constitution characteristics | week 0, week 8, week 12
  The scale classification of the patient's constitution according to Traditional Chinese Medicine theory into nine constitutions. The Constitution in Chinese Medicine Questionnaire (CCMQ) consists of 60 items to classify a person into one or more of nine body constitution types: balanced (8 Items), Qi-deficiency (8 Items), Yang-deficiency (7 Items), Yin-deficiency (8 Items), phlegm-wetness (8 Items), wetness-heat (6 Items), blood-stasis (7 Items), Qi-depression (7 Items), and special diathesis (7 Items). A higher score in the CCMQ scale indicates a higher likelihood of the specific body constitution. The original score is sum up each item's score. The conversion score of constitution characteristics is [(original scores- items)/(items*40]*100. The balanced constitution is the converted score >60 and the rest constitutions' converted scores all < 30. The unbalanced constitution is the converted score ≥40.
Changes in the IWQOL - Lite scale score | week 0, week 8, week 12
  Quality of life was examined using the Impact of Weight on Quality of Life (IWQOL) Kids questionnaire, which has a score range from 0(worst) to 100(best).
Changes in the Emotional and Psychological Assessment scale | week 0, week 8, week 12
  10 item self-report measure of psychological distress with five response categories (none of the time, a little of the time, some of the time, most of the time, all of the time). Scores range from 10 to 50; a higher score indicates more psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongyu Zhou, Professor, Principal Investigator — Hubei Hospital of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided
the data will be published in the form of public papers before January 2022 for public inquiries

REFERENCES:
- [Background] Park BY, Lee MJ, Kim M, Kim SH, Park H. Structural and Functional Brain Connectivity Changes Between People With Abdominal and Non-abdominal Obesity and Their Association With Behaviors of Eating Disorders. Front Neurosci. 2018 Oct 11;12:741. doi: 10.3389/fnins.2018.00741. eCollection 2018. PMID 30364290
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Freisling H, Arnold M, Soerjomataram I, O'Doherty MG, Ordonez-Mena JM, Bamia C, Kampman E, Leitzmann M, Romieu I, Kee F, Tsilidis K, Tjonneland A, Trichopoulou A, Boffetta P, Benetou V, Bueno-de-Mesquita HBA, Huerta JM, Brenner H, Wilsgaard T, Jenab M. Comparison of general obesity and measures of body fat distribution in older adults in relation to cancer risk: meta-analysis of individual participant data of seven prospective cohorts in Europe. Br J Cancer. 2017 May 23;116(11):1486-1497. doi: 10.1038/bjc.2017.106. Epub 2017 Apr 25. PMID 28441380
- [Background] Garvey WT, Mechanick JI, Brett EM, Garber AJ, Hurley DL, Jastreboff AM, Nadolsky K, Pessah-Pollack R, Plodkowski R; Reviewers of the AACE/ACE Obesity Clinical Practice Guidelines. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY COMPREHENSIVE CLINICAL PRACTICE GUIDELINES FOR MEDICAL CARE OF PATIENTS WITH OBESITY. Endocr Pract. 2016 Jul;22 Suppl 3:1-203. doi: 10.4158/EP161365.GL. Epub 2016 May 24. PMID 27219496
- [Background] Dalle Grave R, Calugi S, El Ghoch M. Lifestyle modification in the management of obesity: achievements and challenges. Eat Weight Disord. 2013 Dec;18(4):339-49. doi: 10.1007/s40519-013-0049-4. Epub 2013 Jul 27. PMID 23893662
- [Background] Khera R, Murad MH, Chandar AK, Dulai PS, Wang Z, Prokop LJ, Loomba R, Camilleri M, Singh S. Association of Pharmacological Treatments for Obesity With Weight Loss and Adverse Events: A Systematic Review and Meta-analysis. JAMA. 2016 Jun 14;315(22):2424-34. doi: 10.1001/jama.2016.7602. PMID 27299618
- [Background] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Aminian A, Brethauer SA, Navaneethan SD, Singh RP, Pothier CE, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric Surgery versus Intensive Medical Therapy for Diabetes - 5-Year Outcomes. N Engl J Med. 2017 Feb 16;376(7):641-651. doi: 10.1056/NEJMoa1600869. PMID 28199805
- [Background] Ikramuddin S, Korner J, Lee WJ, Connett JE, Inabnet WB, Billington CJ, Thomas AJ, Leslie DB, Chong K, Jeffery RW, Ahmed L, Vella A, Chuang LM, Bessler M, Sarr MG, Swain JM, Laqua P, Jensen MD, Bantle JP. Roux-en-Y gastric bypass vs intensive medical management for the control of type 2 diabetes, hypertension, and hyperlipidemia: the Diabetes Surgery Study randomized clinical trial. JAMA. 2013 Jun 5;309(21):2240-9. doi: 10.1001/jama.2013.5835. PMID 23736733
- [Background] Reis LO, Favaro WJ, Barreiro GC, de Oliveira LC, Chaim EA, Fregonesi A, Ferreira U. Erectile dysfunction and hormonal imbalance in morbidly obese male is reversed after gastric bypass surgery: a prospective randomized controlled trial. Int J Androl. 2010 Oct 1;33(5):736-44. doi: 10.1111/j.1365-2605.2009.01017.x. Epub 2009 Dec 16. PMID 20039972
- [Background] Gloy VL, Briel M, Bhatt DL, Kashyap SR, Schauer PR, Mingrone G, Bucher HC, Nordmann AJ. Bariatric surgery versus non-surgical treatment for obesity: a systematic review and meta-analysis of randomised controlled trials. BMJ. 2013 Oct 22;347:f5934. doi: 10.1136/bmj.f5934. PMID 24149519
- [Background] Yeh TL, Chen HH, Pai TP, Liu SJ, Wu SL, Sun FJ, Hwang LC. The Effect of Auricular Acupoint Stimulation in Overweight and Obese Adults: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2017;2017:3080547. doi: 10.1155/2017/3080547. Epub 2017 Dec 5. PMID 29358964
- [Background] Tronieri JS, Wadden TA, Walsh OA, Berkowitz RI, Alamuddin N, Gruber K, Leonard S, Chao AM. Effects of liraglutide plus phentermine in adults with obesity following 1 year of treatment by liraglutide alone: A randomized placebo-controlled pilot trial. Metabolism. 2019 Jul;96:83-91. doi: 10.1016/j.metabol.2019.03.005. Epub 2019 Mar 20. PMID 30902750
- [Derived] Wang LH, Huang W, Zhou W, Zhou L, Zhou XL, Zhou P, Yan Y, Zhou ZY, Wang H. Moxibustion combined with characteristic lifestyle intervention of Traditional Chinese Medicine in the treatment of abdominal obesity: A study protocol for a randomized controlled trial. Medicine (Baltimore). 2020 Oct 23;99(43):e22855. doi: 10.1097/MD.0000000000022855. PMID 33120822